CLINICAL TRIAL: NCT07371559
Title: Assessment of Calories in the Diets Using 3D Scanning and a Photographic Method
Brief Title: Assessment of Food Intake Using Both 3D Scanning Method and a Photographic Method
Status: Recruiting | Type: Observational
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Other Study IDs: SIAT-IRB-250215-H0960
Record Dates: First submitted 2025-04-03; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Data Collection
Keywords: food intake; food preference; food energy assessment
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: 21.5≤BMI<25, age between 25-40 years old, 100subjects.
- Superlean: 15<BMI≤18.5, age between 25-40 years old, 100 subjects.

SUMMARY:
This project aims to develop a new and more accurate method to assess energy intake in the diet by collaborating with Astravis company in Switzerland, integrating image recognition and intelligent applications, to improve the accuracy of energy assessment in the food, and to explore the application in dietary research.The researchers will recruit 200 volunteers.

DETAILED DESCRIPTION:
This study will provide food for the participants, and they will independently choose their preferred food for consumption according to their usual dietary habits. This study will take 3D scanning and photography of the food plates before and after eating to analyze the energy intake by each participant.

ELIGIBILITY:
Inclusion Criteria:

Recently measured body mass index (BMI): normal control group (21.5 ≤ BMI < 25); Recently measured body mass index (BMI): healthy underweight group (15 < BMI ≤ 18.5); Must be able to choose the food as requested.

Exclusion Criteria:

Metabolic diseases; Recent weight loss due to various disease causes; Ongoing treatment for weight loss; Eating disorders; Pregnant or lactating women; Infectious diseases such as HIV, Hepatitis; Diabetes mellitus.

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants are healthy, with no metabolic disorder, 22 - 40 years old
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
BMI of the volunteers | This study will take about 1 year and a half to finish, starting from May 1 2025 to Dec 31 2026.
  The volunteers' BMI is chosen between normal and underweight for easy comparison.
3D scanning of the foods chosen by volunteers using a Bodyscan3d smartphone application | This study will take about 1 year and a half to finish, starting from May 1 2025 to Dec 31 2026.
  The volunteers will be asked to choose 5 out of 20 dishes in a buffet and 3D scanning of the foods chosen by volunteers will be taken using a Bodyscan3d application.
Weight and name of each food | This study will take about 1 year and a half to finish, starting from May 1 2025 to Dec 31 2026.
  The weight and name of the food selected by the volunteers will be systematically recorded using a digital electronic scale and food record form. This scale and food record form will be employed to ensure accurate measurements of each food item's mass that the volunteers consume throughout the study period and each food item they choose.
Calories of the food chosen by the volunteers will be evaluated using the Hava smartphone application | This study will take about 1 year and a half to finish, starting from May 1 2025 to Dec 31 2026.
  We use another Hava application to evaluate the calories of the food selected by the volunteers and compare with the calories we calculated, with the smaller the difference, the better the Hava assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Institute of Advanced Technology, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No